CLINICAL TRIAL: NCT04980443
Title: CELTiC Trial: an International Multicentre Study Evaluating the CELTiC Panel for the Detection of Advanced Neoplasia in Fecal Immunochemical Test (FIT)-Positive Individuals
Brief Title: Evaluation of a New Blood-based Test to Detect Colorectal Cancer and Its Precursors
Acronym: CELTiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Bergman Clinics (Other); University of Bologna (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Professor doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NL77730.018.21
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Polyp; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: We will cross-sectionally assess the CELTiC test in a group of FIT-positive individuals.
Masking Description: Endoscopy staff will be blinded to the result of the CELTiC test. Additionally, laboratory staff that assesses the CELTiC test will be blinded to the result of the colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIT positive individuals (Experimental): FIT-positive individuals of whom we will collect blood samples and who will undergo a colonoscopy after blood sampling.
  Interventions: Diagnostic Test: CELTiC test

INTERVENTIONS:
Diagnostic Test: CELTiC test — The CELTiC test is a blood-based test consisting of four mRNA markers and the risk factor age.

SUMMARY:
The CELTiC panel is a potential blood-based test for detecting colorectal cancer (CRC) and precursors of CRC. This can be useful for CRC screening, since this requires tests that detect cancer in an early stage to maximize the chances of successful treatment.

CELTiC combines four markers that can be detected in blood. These markers are composed of so-called messenger RNA (mRNA) and can be viewed as the instructions of our genes to the cell to make certain proteins. Cancer is the result of mutation in these genes. Thus, the mRNA in cancer patients is, depending on the type of mRNA, often abnormal. In earlier studies, the developers of CELTiC found four mRNA's that are different in patients with CRC compared to healthy individuals. However, CELTiC has not yet been extensively studied in individuals for whom the test is intended: a population undergoing CRC screening.

The current study aims to fill this gap. We will assess the ability of CELTiC to detect CRC and precursors of CRC in a population of individuals between 50 and 75 years old in the Netherlands and Italy. This population has already been preselected by having a positive fecal immunochemical test (FIT), a test that is frequently used in CRC screening. This population will undergo a colonoscopy, a procedure where a doctor enters the large bowel through the anus using a flexible camara to assess whether the patient has cancer. Prior to this colonoscopy, we will collect blood samples from the individuals to assess their CELTiC score. After the colonoscopy and the blood analysis, we can assess whether the test adequately detects CRC and precursors of CRC in this population.

DETAILED DESCRIPTION:
1. BACKGROUND

   Colorectal Cancer (CRC) is one of the leading causes of cancer in developed regions around the world and its incidence is rising(1,2). Many nations or regions have introduced CRC population screening programmes to detect cancerous lesions before symptoms arise or to detect precursor lesions whose eradication may prevent CRC (3).

   The Faecal Immunochemical Test (FIT) is used to screen for CRC in many nations and regions around the world. Its advantages include ease of use, the ability to be performed at home and to be sent by mail to a laboratory, and its cost-efficiency (4). Moreover, these characteristics enable population-wide screening without the need for all participants to undergo a colonoscopy.

   However, a downside of the FIT is its performance. In the Netherlands, where a FIT cut-off concentration of 47 mcg Hb/g faeces is used, the FIT produces a negative result in 15% of people who have CRC (5). For the detection of CRC and Advanced Adenomas (AA), referred to as Advanced Neoplasia (AN), the FIT falsely provides a negative result in up to 70% of people with AN. In addition, more than half of the people with a positive FIT result in the Netherlands do not have any (pre)cancerous lesions at colonoscopy.

   One way to improve the efficiency of CRC screening is to introduce a second test to FIT-positive screening participants, to further select individuals for a colonoscopy. Ideally, this test should have a high sensitivity since a false negative result would lead to denying a colonoscopy to a FIT-positive individual with a (pre)cancerous lesion. In addition, the specificity of this test should be high enough to substantially reduce the number of FIT-positive individuals without AN undergoing colonoscopy.

   The CELTiC panel is a blood-based test comprising of four mRNA markers (LGALS4, CEACAM6, TSPAN8, and COL1A2) (6). In a sample of 128 individuals the panel reached an are under the curve (AUC) of 0.82 in discriminating individuals with AN (n = 92; AA n = 25, CRC n = 67) from individuals with a positive FIT result but a normal colonoscopy (n = 36). The CELTiC panel could potentially function as a second test for individuals with a positive FIT result and reduce the number of unnecessary colonoscopies (7). Furthermore, by simultaneously lowering the cut-off concentration of the FIT and introducing the CELTiC panel, screening programs may potentially detect more individuals with AN without increasing the number of colonoscopies performed.
2. QUALITY ASSURANCE

   This cross-sectional diagnostic test study will examine the CELTiC panel in a population of 800 FIT-positive individuals in Italy and the Netherlands. Sites in both nations will adhere to the same protocol, including blood sample collection, processing, and data collection. Monitoring will be put in place at both sites to ascertain adequate data collection and storage. Laboratory personnel and endoscopy staff will be blinded to the results of the colonoscopy and lab analysis respectively.
3. OBJECTIVES

   Primary Objective: to estimate the sensitivity of the CELTiC panel for detecting AN at a cut-off with an expected sensitivity of 90%. Secondary Objective(s) include: (i) to estimate the specificity of the CELTiC panel for detecting AN at a cut-off with an expected sensitivity of 90%; (ii) to estimate the positive predictive value of the CELTiC panel for detecting advanced neoplasia at a pre-specified threshold with an expected sensitivity of 90%; (iii) to estimate the specificity of the CELTiC panel for detecting advanced neoplasia and CRC at an observed sensitivity of 90%; (iv) to estimate the positive predictive value of the CELTiC panel for detecting advanced neoplasia and CRC at on observed sensitivity of 90%; (v) to estimate the Area under the receiver operator characteristic curve (c-statistic); (vi) to estimate the association between CELTiC score and FIT concentration.
4. SAMPLE SIZE

The CRC screening programs of Italy and the Netherlands differ in multiple aspects: in Italy, individuals between 50 and 69 years old are screening every two years with FIT set at a threshold of 20 ug Hb/g feces. In contrast, the Netherlands screens individuals between 55 and 75 years old every two years with FIT set at a threshold of 47 ug Hb/g feces. Therefore, if we were to analyse the results from a combination of these two populations, the results may not be externally valid; the population would consist of more individuals with a relatively high FIT results compared to any other FIT-population in the world. Since FIT is an important risk factor for AN, this may induce selection bias.

Therefore, we have opted to perform two analyses: one with all individuals recruited in Italy (FIT >= 20), and one with all individuals with a FIT of 47 ug Hb/g or higher (both in the Netherlands and Italy). We will aim to estimate a cut-off of CELTiC with a sensitivity of 90% for detecting AN. In addition, we are interested in an estimate with a 95% confidence interval that is not wider than 5% at either side and, for practical reasons, to split the recruiting between Italy in the Netherlands in a 3:2 ratio. Given the positive predictive value of FIT in both screening programs at their respective cut-offs, we will need in total 800 participants for this trial, 347 of whom need to be diagnosed with AN.

ELIGIBILITY:
Inclusion Criteria:

* FIT concentration of 20 ug Hb/g or higher (Italy) or 47 ug Hb/g or higher (Netherlands) in the national CRC screening program as reason for referral.
* Age between 55 and 75 years (Netherlands) or 50 and 69 years (Italy)

Exclusion Criteria:

* No signed informed consent
* History or current treatment for colorectal cancer
* History of inflammatory bowel disease
* History of other condition for which colonoscopy surveillance is planned within the next 5 years.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CELTiC | AN will be measured at colonoscopy, right after the blood samples needed to assess CELTiC have been collected. Analysis of the blood samples will be conducted after colonoscopy.
  The sensitivity of the CELTiC test for detecting advanced neoplasia

SECONDARY OUTCOMES:
Specificity of CELTiC | AN will be measured at colonoscopy, right after the blood samples needed to assess CELTiC have been collected. Analysis of the blood samples will be conducted after colonoscopy.
  The specificity of the CELTiC test
Positive Predictive Value of CELTiC | AN will be measured at colonoscopy, right after the blood samples needed to assess CELTiC have been collected. Analysis of the blood samples will be conducted after colonoscopy.
  The positive predictive value of CELTiC
C-statistic of CELTiC | AN will be measured at colonoscopy, right after the blood samples needed to assess CELTiC have been collected. Analysis of the blood samples will be conducted after colonoscopy.
  The c-statistic of CELTiC for detecting advanced neoplasia

OTHER OUTCOMES:
Association between CELTiC test score and FIT concentration | AN will be measured at colonoscopy, right after the blood samples needed to assess CELTiC have been collected. Analysis of the blood samples will be conducted after colonoscopy. FIT will be collected from the national CRC screening databases.
  Association between CELTiC test score and FIT concentration

CONTACTS AND LOCATIONS:
Locations (4):
- Università di Bologna, Bologna, Emilia-Romagna, Italy
- Netherlands (3):
  - Amsterdam UMC, locatie Academisch Medisch Centrum, Amsterdam, North Holland
  - Bergman Clinics, Amsterdam, North Holland
  - Erasmus University Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Schreuders EH, Ruco A, Rabeneck L, Schoen RE, Sung JJ, Young GP, Kuipers EJ. Colorectal cancer screening: a global overview of existing programmes. Gut. 2015 Oct;64(10):1637-49. doi: 10.1136/gutjnl-2014-309086. Epub 2015 Jun 3. PMID 26041752
- [Background] Ran T, Cheng CY, Misselwitz B, Brenner H, Ubels J, Schlander M. Cost-Effectiveness of Colorectal Cancer Screening Strategies-A Systematic Review. Clin Gastroenterol Hepatol. 2019 Sep;17(10):1969-1981.e15. doi: 10.1016/j.cgh.2019.01.014. Epub 2019 Jan 16. PMID 30659991
- [Background] Rodia MT, Solmi R, Pasini F, Nardi E, Mattei G, Ugolini G, Ricciardiello L, Strippoli P, Miglio R, Lauriola M. LGALS4, CEACAM6, TSPAN8, and COL1A2: Blood Markers for Colorectal Cancer-Validation in a Cohort of Subjects With Positive Fecal Immunochemical Test Result. Clin Colorectal Cancer. 2018 Jun;17(2):e217-e228. doi: 10.1016/j.clcc.2017.12.002. Epub 2017 Dec 12. PMID 29352642
- [Background] Ferlizza E, Solmi R, Miglio R, Nardi E, Mattei G, Sgarzi M, Lauriola M. Colorectal cancer screening: Assessment of CEACAM6, LGALS4, TSPAN8 and COL1A2 as blood markers in faecal immunochemical test negative subjects. J Adv Res. 2020 Mar 3;24:99-107. doi: 10.1016/j.jare.2020.03.001. eCollection 2020 Jul. PMID 32257432
- [Background] Senore C, Basu P, Anttila A, Ponti A, Tomatis M, Vale DB, Ronco G, Soerjomataram I, Primic-Zakelj M, Riggi E, Dillner J, Elfstrom MK, Lonnberg S, Sankaranarayanan R, Segnan N. Performance of colorectal cancer screening in the European Union Member States: data from the second European screening report. Gut. 2019 Jul;68(7):1232-1244. doi: 10.1136/gutjnl-2018-317293. Epub 2018 Dec 10. PMID 30530530
- [Background] Rodia MT, Ugolini G, Mattei G, Montroni I, Zattoni D, Ghignone F, Veronese G, Marisi G, Lauriola M, Strippoli P, Solmi R. Systematic large-scale meta-analysis identifies a panel of two mRNAs as blood biomarkers for colorectal cancer detection. Oncotarget. 2016 May 24;7(21):30295-306. doi: 10.18632/oncotarget.8108. PMID 26993598
- [Derived] Kortlever TL, Ferlizza E, Lauriola M, Borrelli F, Porro A, Spaander MCW, Bossuyt PM, Ricciardiello L, Dekker E. Diagnostic Accuracy of an Add-On, Blood-Based Screening Test for Colorectal Cancer in Two Established Screening Programmes. Aliment Pharmacol Ther. 2025 Jun;61(12):1935-1943. doi: 10.1111/apt.70141. Epub 2025 Apr 10. PMID 40207404